CLINICAL TRIAL: NCT06479044
Title: Application Of Herrmann's Brain Quadrant Model and Its Relationship With Learning Styles in Anesthesiology Residents
Brief Title: Applying Herrmann's Brain Quadrant Model to Learning Styles in Anesthesiology Residents
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Clotilde Fuentes-Orozco, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: Herrmann's Brain Quadrant
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Learning Problem
Keywords: Residency; Learning; Herrmann´s Model; Medical Knowledge; Cognitive Function

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- LC- Scientific Expert
  Interventions: Diagnostic Test: Herrmann Brain Model
- LL- Organizer-Introvert
  Interventions: Diagnostic Test: Herrmann Brain Model
- RC- Interpersonal Strategist
  Interventions: Diagnostic Test: Herrmann Brain Model
- RL- Imaginative Communicator
  Interventions: Diagnostic Test: Herrmann Brain Model

INTERVENTIONS:
Diagnostic Test: Herrmann Brain Model — The test comprises 120 multiple-choice items on academic, daily, and professional scenarios

SUMMARY:
the ability to learn and adapt to clinical demands is essential in the training of residents. The Herrmann Brain Model categorizes thinking styles based on the preference for utilizing brain quadrants, serving as an applied tool for residents to assess their learning preferences.

DETAILED DESCRIPTION:
This study delineates the learning styles according to Herrmann's brain quadrant model among anesthesiology residents at the National Western Specialty Hospital, Mexican Social Security Institute. Cross-sectional descriptive study; the Herrmann Brain Dominance Test was administered to anesthesiology residents. Each brain quadrant embodies distinct characteristics, thinking patterns, and approaches to knowledge acquisition. The test comprises 120 multiple-choice items on academic, daily, and professional scenarios. The quadrants are described as follows: LC "Scientific Expert," LL "Organizer-Introvert," RC "Interpersonal Strategist," RL "Imaginative Communicator."

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology residents of the National Western Specialty Hospital, Mexican Social Security Institute

Exclusion Criteria:

* Residents of other specialties of the National Western Specialty Hospital, Mexican Social Security Institute

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Physicians between 27 and 32 years of age of both genders
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Quadrant dominance | 12 months
  Determine the learning style of each one of them based on the predominant cerebral hemisphere

CONTACTS AND LOCATIONS:
Locations (1):
- National Western Speciality Hospital, Mexican Social Security Institute, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No